CLINICAL TRIAL: NCT06123832
Title: Study of the Clinical Benefits of Different Formulations of Amphotericin B
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Qianfoshan Hospital (Other)
Responsible Party: Principal Investigator, Rui Yang, Associate professor of pharmacy, Qianfoshan Hospital
Other Study IDs: LCYX-YR-20230102
Record Dates: First submitted 2023-11-03; First posted 2023-11-09 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2023-11

CONDITIONS: Efficacy; Safety
Keywords: Liposomal Amphotericin B for Injection; Amphotericin B Cholesteryl Sulfate Complex for Injection; Amphotericin B for Injection; Safety; Efficacy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Experimental Group: Liposomal Amphotericin B for Injection (Ampicillin®)
- Control Group: Liposome of Amphotericin B for Injection (Fungoxone®), Cholesteryl Sulfate Complex of Amphotericin B for Injection (Amphotericin®), Amphotericin B for Injection

SUMMARY:
This project intends to carry out a multi-center retrospective observational real-world study to understand the current status of amphotericin B use by formulation type, compare the differences in safety and efficacy of each formulation in domestic clinical application, provide real-world evidence for clinical drug selection, and provide evidence-based evidence in support of rational clinical drug use.

DETAILED DESCRIPTION:
The researchers selected patients with amphotericin B use records discharged from five tertiary hospitals across the country from January 1, 2020 to the present, extracted data according to the inclusion and exclusion criteria, and divided them into experimental and control groups, in order to understand the current status of amphotericin B use in each preparation type, compare the differences in the safety and efficacy of the various preparations in the domestic clinical application, and provide real-world evidence of the choice of clinical medication.

ELIGIBILITY:
Inclusion Criteria:

1. Patients discharged from January 1, 2020 to the present;
2. Patients with a record of amphotericin B use.

Exclusion Criteria:

1.Key information missing from patient studies.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with documented amphotericin B use discharged from 5 tertiary care hospitals across the country from January 1, 2020 to the present were selected for the study to exclude patients with missing key information for the study and were divided into experimental and control groups for the study.
Sampling Method: Non-Probability Sample
Enrollment: 184 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall Adverse Reaction Rate | Through study completion,up to half a year.
  The incidence of total adverse reactions was analyzed to assess the difference in safety of amphotericin B by formulation type in domestic clinical application, to provide real-world evidence for clinical drug selection, and to provide evidence-based evidence in support of rational clinical drug use.
Pathogen clearance rate | Through study completion,up to half a year.
  To assess the differences in effectiveness of amphotericin B by formulation type in domestic clinical application by analyzing the pathogen clearance rate, to provide real-world evidence for clinical dosing selection, and to provide evidence-based evidence to support rational clinical dosing.

CONTACTS AND LOCATIONS:
Overall Officials: Rui Yang, MD, Principal Investigator — Qianfoshan Hospital
Locations (1):
- Rui Yang,MD, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No